CLINICAL TRIAL: NCT03837626
Title: Estrogen Receptor Alpha Signaling in Endothelial Cells Exacerbates Arterial Stiffening Via Upregulation of ENaC in Insulin Resistant Females
Brief Title: ENAC Blockade and Arterial Stiffness
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Camila Manrique, MD, Associate Professor, Endocrinology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012990
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Overweight and Obesity; Insulin Resistance
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance | interventions — Amiloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): 6 months of daily placebo
  Interventions: Drug: Placebo - Cap
- Amiloride (Experimental): 6 months of amiloride (max dose 5 mg) treatment
  Interventions: Drug: Amiloride Pill

INTERVENTIONS:
Drug: Placebo - Cap — 6 months of 1 pill a day
  Arms: Placebo
Drug: Amiloride Pill — Max dose of 5 mg a day for 6 months
  Arms: Amiloride

SUMMARY:
To determine whether treatment with the ENaC inhibitor, amiloride, improves endothelial function and arterial stiffness in obese insulin resistant subjects in a randomized placebo-controlled trial examining pre and postmenopausal women and age-matched men.

DETAILED DESCRIPTION:
Overweight/obese males, pre- and post-menopausal females with insulin resistance, 30-70 years of age will be recruited. Following screening, eligible men and women will be randomly assigned to either amiloride (max dose 5mg) or placebo in a double-blinded design manner.

After randomization, subjects will be scheduled for an outpatient visit to the undergo baseline assessment of arterial stiffness (carotid femoral pulse wave velocity - cfPWV) and endothelial function (brachial popliteal artery flow mediated dilation). Subject assessment will be repeated at 12 weeks and at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 70 years of age at randomization
* Body mass index (BMI) 25.1-50 kg/m2 or waist circumference > 88 cm (> 35 in) in women and >102 cm (>40 in) in men. 3, 4
* One other characteristic of metabolic syndrome (elevated triglycerides ≥150 mg/dl; HDL cholesterol <40 mg/dl in men and <50 mg/dl in women; blood pressure ≥130/85 mm Hg or treatment for hypertension; impaired fasting glucose (≥100 mg/dl)) or fasting insulin level >10 mU/L (correlates with insulin resistance).

Exclusion Criteria:

1. History of type 1 or type 2 diabetes
2. Known cardiovascular events within the last 12 months (stroke, acute coronary event, revascularization, heart failure hospitalization).
3. History of uncontrolled thyroid disease, chronic liver disease (cirrhosis) or GFR <50 ml/min.
4. Use of potassium sparing medications (angiotensin II receptor blockers, angiotensin converting enzymes inhibitors or mineralocorticoid receptor blockers) or use of potassium supplements.
5. Active cancer (This criterion does not apply to those subjects with basal cell carcinoma or stage 1 squamous cell carcinoma of the skin)
6. Excessive alcohol consumption (>14 drinks/week for men, >7 drinks/week for women)
7. Current tobacco use
8. Non controlled hypertension
9. Participation in regular exercise > 3 days/wk per week at a moderate or vigorous intensity
10. Pregnancy or lactation in women (or women not using contraceptives)
11. Women who plan to become pregnant during the duration of the trial
12. Chronic use of NSAIDs
13. Potassium level > 5.0 mqE/L at time of screening
14. Blood pressure at screening <110/70

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camila Manrique Acevedo, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Amiloride
Started | 47 | 90
Completed | 37 | 79
Not Completed | 10 | 11
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 2 | 3
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Amiloride | Total
Number analyzed (Participants) | 47 | 90 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 86 | 128
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 59 | 87
  Male | 19 | 31 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 44 | 87 | 131
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 40 | 80 | 120
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 90 | 137

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Systolic blood pressure obtained during experimental visits at the different time points
Time Frame: 3 and 6 mo
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Amiloride
Number analyzed (Participants) | 37 | 79
mmHg
  3 mo | 127.53 [123.07 to 132] | 122.90 [119.85 to 125.94]
  6 mo | 125.51 [121.11 to 129.92] | 120.27 [117.25 to 123.30]

2. Other Pre Specified Outcome: Brachial Artery Flow Mediated Dilation (FMD)
Description: Brachial artery flow-mediated dilation will be assessed at baseline, 12, and 24 weeks. FMD is a measurement of conduit artery endothelial function.
Time Frame: Baseline, 3 months (interim) and 6 months (final)
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | Amiloride
Number analyzed (Participants) | 32 | 70
Percentage
  3 months (interim) | 6.03 (0.62) [4.90 to 7.17] | 6.25 (0.42) [5.49 to 7.02]
  Delta 6 months (final) | 5.59 (0.56) [4.50 to 6.68] | 6.16 (0.44) [5.42 to 6.90]

3. Other Pre Specified Outcome: Popliteal Artery Flow Mediated Dilation (FMD)
Description: Popliteal artery flow-mediated dilation will be assessed at baseline, 12, and 24 weeks. FMD is a measurement of conduit artery endothelial function.
Time Frame: Baseline, 3 months (interim) and 6 months (final)
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | Amiloride
Number analyzed (Participants) | 14 | 34
Percentage
  3 months (interim) | 1.71 (0.30) [0.74 to 2.69] | 2.22 (0.29) [1.59 to 2.84]
  6 months (final) | 1.80 (0.31) [0.91 to 2.69] | 2.55 (0.34) [2.02 to 3.09]

4. Primary Outcome: Carotid Femoral Pulse Wave Velocity
Description: cfPWV is the gold standard of arterial stiffness. It was assessd during experimental visits, under the same conditions in a blinded manner
Time Frame: baseline, 3 and 6 mo
Population: Number of participants that finished clinical trial
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Placebo | Amiloride
Number analyzed (Participants) | 37 | 97
m/s
  3 months | 7.25 [6.85 to 7.65] | 6.80 [6.53 to 7.07]
  6 months | 7.12 [6.73 to 7.51] | 6.81 [6.54 to 7.08]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Amiloride
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/90
Other Adverse Events (participants affected / at risk) | 5/47 | 9/90
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Amiloride (N=90)
Headache (Nervous system disorders) | 5 (5) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03837626/Prot_001.pdf
  • Statistical Analysis Plan (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT03837626/SAP_003.pdf
  • Informed Consent Form (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03837626/ICF_000.pdf